CLINICAL TRIAL: NCT02456298
Title: Comparing Behavioral Assessments Using Telehealth for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew J O'Brien, PhD, BCBA-D (Other)
Collaborators: University of Houston (Other); Emory University (Other); Children's Healthcare of Atlanta (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Matthew J O'Brien, PhD, BCBA-D, Clinical Psychologist/Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#201501781; R01MH104363 (NIH)
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Telehealth; Applied behavior analysis
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard FA+FCT (Active Comparator): Parents are coached via weekly telehealth visits to use Functional Analysis (FA) to assess problem behavior and Functional Communication Training (FCT) to treat the problem behavior identified.
  Interventions: Behavioral: Standard FA+FCT
- Pragmatic FA+FCT (Experimental): Parents are coached via weekly telehealth visits to use a brief, streamlined version of Functional Analysis (FA) to assess problem behavior and to follow that assessment with Functional Communication Training (FCT) to treat the problem behavior identified. The version of FCT used in the Pragmatic arm involves significantly less data scoring and graphing than the version used in the Standard arm.
  Interventions: Behavioral: Pragmatic FA+FCT

INTERVENTIONS:
Behavioral: Standard FA+FCT — Standard Functional Analysis and Functional Communication Training
  Arms: Standard FA+FCT
Behavioral: Pragmatic FA+FCT — Pragmatic Functional Analysis and Functional Communication Training
  Arms: Pragmatic FA+FCT

SUMMARY:
The main purpose of this study is to determine the most efficient way for families to reduce problem behavior in their children with an autism spectrum disorder. Parents will be trained using telehealth to use applied behavior analysis (ABA) procedures to improve child behavior and communication. The study compares an established type of ABA assessment and treatment to a briefer, more streamlined version of this same type of assessment/treatment.

DETAILED DESCRIPTION:
Managing challenging behavior in autism spectrum disorders (ASD) can profoundly improve quality of life for children and families. However, many families lack access to research-based treatment, such as applied behavior analysis (ABA). This study is a randomized trial comparing outcomes of treatment for ASD using either a standard Functional Analysis Plus Functional Communication Training (FA+FCT) package or a pragmatic version that offers a briefer, less time-intensive model of FA+FCT. Both types of FA+FCT are provided via telehealth in family homes to maximize generalizability to real-life settings. Providing ABA through telehealth makes an effective treatment accessible across geographic barriers so that no child is excluded based on where they live. The study also examines key family factors that influence successful outcomes.

The study has 3 primary aims: (1) To assess outcomes for ABA telehealth by assigning children to either a Pragmatic FA+FCT group or to a group receiving Standard FA+FCT. Outcomes will be compared based on the percent reduction in problem behavior, communication increases, time to achieve outcomes, treatment fidelity, family acceptance of treatment, and generalization and maintenance of treatment gains. (2) The study will assess the relation of family factors to treatment efficacy and acceptability by assessing parent stress, mood, and social support in relation to outcomes. (3) Cost effectiveness will be assessed in relation to the treatment methods used and the efficiency of ABA telehealth.

The study will include 102 children who meet eligibility criteria from among a larger sample of 150 children. Thirty-six children will receive intervention in each of three states: Iowa, Georgia, and Texas. Study design is a randomized trial using an intent-to-treat analysis. Half of the sample will be randomized to Pragmatic FA+FCT and half to Standard FA+FCT. Treatment will be provided via telehealth using FCT, which is a function-based ABA technique in which parents are trained to be therapists under the direction of behavior consultants. Study procedures typically are completed within 6 months, and follow-up assessments occur 6 months after treatment completion. Data analyses include comparisons between assessment groups, single-case designs examining responses in individual children, cost analyses, and regression analyses of the effects of family factors on outcomes.

The investigators prior research shows that problem behavior can be reduced by over 90% in most children with ASD after 4-6 months of telehealth treatment. If Pragmatic FA+FCT can reduce problem behavior at rates comparable to Standard FA+FCT, then treatment can be started sooner and families can achieve successful outcomes at lower cost. Although pragmatic FA+FCT provides less behavioral information, it may be more resistant to treatment relapse because it does not involve reinforcing high rates of problem behavior.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of autism spectrum disorder
* Significant behavior problems requiring treatment
* At least one parent willing to be trained in behavior analysis via telehealth

Exclusion Criteria:

* Unstable or degenerative neurological disorder

Ages: 18 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2015-06; Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Percent Reduction in Problem Behavior | Change from Baseline to End of Treatment (typically within 4-6 mos.)
  Rate of problem behavior (destruction, aggression, self-injury, noncompliance, etc.) is computed by scoring the frequency of these target behaviors during observation sessions completed before treatment and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J O'Brien, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data for individual participants will be made available through the National Database for Autism Research (NDAR) using the access tools and procedures implemented within NDAR. NDAR is one of the databases that is part of the NIMH Data Archive.
Supporting Information: CSR
Time Frame: Descriptive data will be available as soon as the study has been completed and data have been entered in NDAR. Experimental data will not be available until all treatment and follow-up data have been completed and the initial publications for the study have been published.
Access Criteria: Access criteria are established by NDAR. Additional information about data access for scientists can be obtained at the URL listed below.
URL: https://nda.nih.gov/